CLINICAL TRIAL: NCT01971528
Title: Central and Peripheral Fatigue in Individuals With Parkinson's Disease - Evaluation and Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Associate Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100-3167A3
Record Dates: First submitted 2013-10-18; First posted 2013-10-29 (Estimated); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease(PD)
Keywords: Muscle strength, fatigue, electromyography (EMG), central fatigue, strength straining
MeSH Terms: conditions — Parkinson Disease; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Stage 1: Health control (No Intervention): pilot study: Establishing the central and peripheral contributing factors to the voluntary muscle strength loss during a fatiguing exercise in young and PD groups.
- Stage 1: PD subjects (No Intervention): pilot study: Establishing the central and peripheral contributing factors to the voluntary muscle strength loss during a fatiguing exercise in young and PD groups.
- Stage 2: Health subjects (No Intervention): pilot study: Finding optimal sensory stimulation parameters for PD individuals.
- Stage 2: PD subjects (No Intervention): pilot study: Finding optimal sensory stimulation parameters for PD individuals.
- Stage 3: PD subjects (Experimental): Investigating the long-term effects of combined sensory stimulating strengthening program on the activation level and central fatigue in PD individuals.
  Interventions: Device: Electronic muscle stimulator; Other: Muscle strength training
- Stage 3: PD subjects (Control Subjects) (No Intervention): Investigating the long-term effects of combined sensory stimulating strengthening program on the activation level and central fatigue in PD individuals.

INTERVENTIONS:
Device: Electronic muscle stimulator — Participants will perform 8 weeks of electrical stimulation for Quadriceps muscle belly(30 minutes/time, 3 times/week).
  Arms: Stage 3: PD subjects
Other: Muscle strength training — Participants will perform 8 weeks of isotonic contraction muscle strength training for lower extremities.
  Arms: Stage 3: PD subjects

SUMMARY:
Fatigue is one of the most common symptoms in individuals with Parkinson's Disease (PD). Past research indicated that more than half of the individuals with PD demonstrated fatigue symptom. The severity of fatigue was also correlated to the quality of life in individuals with PD. Finding the contributions of the central and the peripheral factors to fatigue and developing an effective training program for individuals with PD are very important.

Fatigue can be categorized into peripheral or central causes. The central fatigue and voluntary activation failure originate from the decrease in motivation or the reduction of the conduction within corticospinal tracts. Long term activation failure and central fatigue will cause disuse of muscle and result in peripheral weakness and peripheral fatigue. Quantifying the weighting of central versus peripheral factors contributing to the fatigue in people with PD is important.

Most of the conventional strength and endurance training programs were based on the researches of young groups. Almost no training program was design for enhancing the voluntary activation level and relief the central fatigue. Seeking an appropriate training program to enhance central activation is very important for individuals with PD who prone to fatigue.

Previous studies have shown that increasing afferent input by peripheral electrical stimulation (ES) at sensory threshold enhanced the plasticity of contralateral primary sensory cortex, the excitability of corticospinal tracts, and the functional performance in young adults. Combining afferent input with strength training was more effective than strength training along. ES, which is easy to quantify the dose of afferent input, is a feasible method to provide such training.

The purpose of this project is to investigate the effects of the combination of ES at sensory threshold and strength training on voluntary activation in the individuals with PD.

ELIGIBILITY:
Health subjects:

Exclusion Criteria:

* Musculoskeletal injuries for knee.
* Osteoporosis.
* Diabetes.

PD subjects:

Inclusion Criteria:

* Clinical diagnosis of Parkinson disease.

Exclusion Criteria:

* Musculoskeletal injuries for knee.
* Osteoporosis.
* Diabetes.
* Any peripheral or central nervous system injury or disease patients.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-12-18 (Actual); Primary Completion 2014-09-11 (Actual); Study Completion 2015-05-10 (Actual)

PRIMARY OUTCOMES:
Muscle twitch force | baseline, 8 weeks.
  Measure of changes in muscle twitch force by interpolation twitch technique.
Muscle voluntary activity level | Baseline,8 weeks
  Measure of changes in muscle voluntary activity level by interpolation twitch technique.
Muscle strength test for lower extremities. | Baseline, 8 weeks
  Measure of changes in muscle strength test by clinical test.
The central activation and the excitability of motor cortex | Baseline,8 weeks
  Measure of changes in the central activation and the excitability of motor cortex by Transcranial magnetic stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan